CLINICAL TRIAL: NCT06584682
Title: Effects of Sub-occipital Muscle Inhibition Technique on Hamstring Flexibility in Post-laminectomy Patients
Brief Title: Effects of Sub Occipital Muscle Inhibition Technique on Hamstring Flexibility in Post-laminectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01935 Safia Gul
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hamstring Tightness
Keywords: Sub-occipital muscle inhibition technique; cervical traction; muscle energy technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-occipital muscle inhibition technique (Experimental): Therapist puts finger pads just beneath the superior nuchal line (below the occiput and above the C2 vertebra), and lifts the patient head slightly and apply an anterior force with cephalic traction on cervical spine this area. Then straighten the fingers to press the finger tips into muscle and hold until relaxation(30 sec) and then drop the head into palm in new position, give this technique in 10 rep/2 sets (each set have 5 repetitions).hot packs for 15 minutes prior to session, cervical muscle stretching,cervical mechanical traction for 8-10 minutes, force is applied 1/6th of the patient body weight, for C1-C2 at 0 degree of cervical flexion and for below C2 at 20 degree of cervical spine flexion. and cervical muscle Muscle Energy Techniques.
  Interventions: Other: Sub-occipital muscle inhibition technique
- conventional therapy (Other): stretching of hamstring muscle, METs, sciatic nerve glides, lower limb neurodynamic.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Sub-occipital muscle inhibition technique — Therapist puts finger pads just beneath the superior nuchal line (below the occiput and above the C2 vertebra), and lifts the patient head slightly and apply an anterior force with cephalic traction on cervical spine this area. Then straighten the fingers to press the finger tips into muscle and hold until relaxation(30 sec) and then drop the head into palm in new position, give this technique in 10 rep/2 sets (each set have 5 repetitions).hot packs for 15 minutes prior to session, cervical muscle stretching,cervical mechanical traction for 8-10 minutes, force is applied 1/6th of the patient body weight, for C1-C2 at 0 degree of cervical flexion and for below C2 at 20 degree of cervical spine flexion and cervical muscle METs
  Arms: Sub-occipital muscle inhibition technique
Other: conventional therapy — stretching of hamstring muscle, METs, sciatic nerve glides, lower limb neurodynamics.
  Arms: conventional therapy

SUMMARY:
to find out the effects of sub-occipital muscle inhibition technique in combination with upper cervical spine exercises on hamstring muscle flexibility in post-laminectomy patients.

DETAILED DESCRIPTION:
Laminectomy is a decompression surgery which is performed to decrease pressure on spinal nerves. In this surgical procedure a small bone of vertebrae called lamina is removed. Hamstring muscle stiffness is a major problem in post-laminectomy patients, which results in chronic pain, functional limitation and affect patients activity of daily life.

In post-laminectomy patients hamstring stiffness is more profound than iliotibial Band and piriformis stiffness. Sub-occipital muscle and hamstring are connected via a single neural pathway called superior back line which passes through dura matter. Dura matter is the outer most covering of meninges, Sub Occipital Muscles attached to dura matter by Myodural Bridge through vertebral dural ligament. This connection provides a window for relaxation of dural fascia to decrease tone of connected muscular-skeletal units (in which hamstring is also included). So if any of these muscle units become tight, or tone deterioration occur the other unit is automatically malfunctioned. The study shows that if tone sub-occipital muscle falls, it has been reported that the tone of knee flexors such as hamstring also decreases due to relaxation of myofascia.

However, in post-laminectomy patients, incorporating a neural pathway connection technique involving sub-occipital muscle inhibition for upper neural pathway Dura release may offer more effective and immediate results on hamstring muscle flexibility in the lower neural pathway The sub-occipital muscle inhibition technique is a method of inducing relaxation of the fascia by applying soft pressure to the sub-occipital area.

The rationale of the present study is to find out the effectiveness of Sub Occipital Muscle inhibition technique for stiff hamstring muscle in post-laminectomy patients, pain and disability. To compare the effectiveness of SOM inhibition technique in combination of upper cervical spine muscle stretching,traction etc. with hamstring muscle stretching, lower limb neurodynamic etc.

ELIGIBILITY:
Inclusion Criteria:

* Hamstring muscle tightness, (AKE < 80) or (more than 20 degree lag in knee extension).
* Back of the thigh pain.
* Prior laminectomy surgical procedure at lumber spine.
* Patients who are willing to participate.

Exclusion Criteria:

* Prior femur and back related fracture,
* Bilateral lower limb pain,
* Any systemic issue.
* Visual hamstring swelling.
* Individual with cervical ligaments instability and migraine.
* Unable to understand the consent form,
* Patients who are not willing to participate in procedure

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Active knee extension test | two weeks
  Patient is supine, unaffected limb on support surface and the examined limb elevated so that hip in 90 degree of flexion and knee to extended position perpendicular to ground. A lag of 20 degrees is considered normal from full extension, less than 20 degrees is considered as hamstring muscle tightness
Numeric pain rating scale | two weeks
  The NPRS is a self-reported, or clinician administered, measurement tool consisting of a numerical point scale with extreme anchors of 'no pain' to 'extreme pain'. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form.
Modified Oswestry disability index | two weeks
  The Oswestry Disability Index (aka the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. There are 10 questions, for each question there is a possible 5 points; 0 for the first answer, 1 for the second answer, etc.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Health and wellness rehabilitation center, Swābi, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No